CLINICAL TRIAL: NCT03624829
Title: Shared Care and Usual Health Care for Mental and Comorbid Health Problems. A Cluster Randomized Trial
Brief Title: Shared Care and Usual Health Care for Mental and Comorbid Health Problems
Status: Completed | Type: Observational
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Torleif Ruud, Senior Researcher, Professor emeritus, University Hospital, Akershus
Other Study IDs: 273932
Record Dates: First submitted 2018-08-05; First posted 2018-08-10 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exp: Patients of GPs with shared care: All patients 16-65 years old who during 12 months have been in contact with a GP in any of the three GP centers that are randomized to shared care before the 12 months.
  Interventions: Other: Shared care
- Con: Patients of GPs without shared care: All patients 16-65 years old who during 12 months have been in contact with a GP in any of the three GP centers that are not randomized to shared care before the 12 months, and all patients 16-65 years old who during 12 months have been in contact with a GP in any of the six GP center before the randomization and implementation of shared care.

INTERVENTIONS:
Other: Shared care — The intervention is an adapted version of shared care with close collaboration by services and professional groups, mainly localized in three GP centers. At each GP center one clinical psychologist specialist from the community mental health center (CMHC) works two and a half day a week, and a psychiatrist from the CMHC work at each GP center 1-2 hours a week. The psychologist and the psychiatrist are available for the GPs for consultation and discussions, and they give assessments and brief treatments to patients as requested by the GPs. Other primary health and social care and other specialized mental health or substance addiction services are involved or consulted according to needs of the patients.
  Groups: Exp: Patients of GPs with shared care

SUMMARY:
The aim is to study the impact on patients and health care by an adaption of the Hamilton Family Health Team model of shared care between general practitioners (GPs), mental health services and other primary or specialized services. The study is done at six GP centers with 30 GPs in three boroughs in Oslo, Norway.

At each GP center with shared care one clinical psychologist from a CMHC works two and a half day a week and a psychiatrist 1-2 hours a week. They are available for the GPs for discussions, and they give assessment and brief treatment as requested by the GPs. Other primary health and social care and other specialized mental health or substance addiction services are consulted according to needs of the patients.

The study is a cluster randomized controlled study of GP patients and their health care in GP centers with shared care (experimental group) compared with usual health care in other GP centers (control group). In each of three boroughs one GP center is randomized to shared care for 18 months while another center continues with usual health care.

Register data on patients and services are extracted for 12 months (T0) before implementation of shared care and for 12 months (T1) with shared care after 6 months implementation. The register data on patients and health care are extracted from the GP patient records, mental health and substance abuse services, and NAV (social/welfare services). The cohorts at T0 and T2 include all patients 16-65 years old seen by the GPs.

Patient-reported mental health, functional impairment due to health problems, overall quality of life and satisfaction with health services are studied for a sub-sample of the register cohort at both T0 and T1.

A qualitative sub-study of experiences with collaboration, the shared care model, implementation of the model, facilitators and barriers is done at the end of the 18 months period of shared care. The informants include patients, GPs and coworkers, and managers and professionals involved with shared care.

The study protocol was approved by the regional and national committees on medical and health research, as well as by the data protection officer at health trust.

Progress and status are described in Detailed description. Data analysis starts in September 2018.

DETAILED DESCRIPTION:
BACKGROUND

There have been various forms of collaboration in Norway between community mental health centres (CMHCs), GPs and primary health and social care. But with a lack of research on such models, there is little knowledge on whether they contribute to better health care, outcome and satisfaction, e.g. for the large group of patients with moderately severe mental and comorbid health problems mostly seen by GPs. There is a great need for clearly defined collaboration models and for research-based knowledge of their feasibility and impact in the context of the Norwegian health services.

Reviews of studies on collaboration show inconsistent results, including insufficient evidence to demonstrate significant benefits from shared care (Smith 2009), modest reductions in primary care consultations and mental health referrals (Harkness 2009), partly improved depression management (Butler 2011), and research primarily on simpler models of collaboration between two professionals (Hviding et al. 2008, Craven et al 2006).

The Family Health Teams model developed in Hamilton, Canada, is a promising model of shared care (Kates 2011a, 2011b). It is built around GP practices. Each team include one or more GPs, nurses, mental health counsellors, a visiting consultant psychiatrist, and some other part-time staff (pharmacist, nutritionist, physiotherapist, occupational therapist). The model has increased access to care for persons with mental health and addiction problems, reduced waiting time, reduced referrals to outpatient mental health services, increased patient satisfaction, improved patient health, improved communication and co-ordination, and increased GPs' confidence and skills in treating mental health problems.

CONTEXT

The study is done in three Oslo boroughs (Alna, Grorud, Stovner) with a total population of 108 000. They are served by a total of 85 GPs in GP centers, by the primary health and social care in the boroughs, and by a community mental health center (CMHC), child and adolescent mental health services (CAMHS) and other departments of the Division Mental Health Services at Akershus University Hospital.

INTERVENTION

The intervention is an adapted version of shared care with close collaboration by services and professional groups, mainly localized in three GP centers. At each GP center one clinical psychologist specialist from the community mental health center (CMHC) works two and a half day a week, and a psychiatrist from the CMHC work at each GP center 1-2 hours a week. The psychologist and the psychiatrist are available for the GPs for consultation and discussions, and they give assessment and brief treatment to patients as requested by the GPs. Other primary health and social care and other specialized mental health or substance addiction services are involved or consulted according to needs of the patients.

The decisions on the adaption of the model were taken by the collaborating services themselves in October-December 2015 after a joint visit to Hamilton by 14 persons and with input from the research group. This secured that the services had ownership and commitment to the model and contributed to make it feasible and useful.

The shared care in the three experimental GP centers was established during the winter of 2016 and were operational for 18 months from the April/May 2016 to October/November 2017. The implementation was supported by discussions in monthly meetings at each GP center for the professionals collaborating on shared care there, and in monthly meetings at the CMHC between the psychologists and psychiatrists in shared care, managers at the CMHC and the principal investigator of the research study.

AIMS

The aim is to study the impact of a Norwegian adaption of the Hamilton Family Health Team model of shared care between general practitioners (GPs), mental health services and other primary or specialised services.

RESEARCH QUESTIONS

1. What are the characteristics of patients seen in the usual GP practices (ICPC-2 codes, mental health problems, comorbidity of mental and somatic health problems)?
2. How is the total usual health care for the GP patients from GPs, primary health and social care, and mental health and substance addiction services?
3. How is the patient-reported mental health, functioning and satisfaction with health services and collaboration in among patients seen in usual GP practices?
4. Is shared care associated with changes in access to mental health care, referrals to specialized mental health care, use of health services and distribution of patients across services?
5. What is the patient course and outcome (waiting time, sick leave, mental health, functioning, duration of treatment) with shared care compared to usual health care?
6. Is there a more integrated care for comorbidity (concurrent mental/somatic/substance addiction problems) in shared care than in usual health care?
7. How are the GP patients' experiences with shared care compared to usual health care?
8. What do health professionals in shared care experience as main advantages and disadvantages of shared care?
9. What do health professionals in shared care identify as facilitating factors or barriers for implementing shared care?

METHODS

CLUSTER RANDOMIZED CONTROLLED REGISTER STUDY ON IMPACT OF SHARED CARE

The study is a cluster randomized controlled study of GP patients and their health care in shared care (experimental group) compared with usual health care (control group). In each of three boroughs one GP center is randomized to have shared care for 18 months while another GP center continues with usual health care. Register data on patients and health care are extracted for 12 months (T0) before the implementation of shared care and for 12 months (T1) with shared care (after 6 months with implementation of the shared care model).

Retrospective register data on patients and use of services for the two 12 months periods (T0 and T1) are extracted from the GP patient records, Akershus University Hospital (mental health and substance addiction services for adults and youth), and NAV (social/welfare services). Patient cohorts at T0 and T1 include all patients 16-65 years old seen by the 30 GPs in 12 months. Based on earlier studies each cohort was expected to be 20-25 000 patients. In 2014 the 30 GPs referred 840 patients to outpatient mental health clinics and 190 to inpatient mental health wards. Based on this, significant changes in referrals to outpatient clinics (main primary outcome) are expected to be shown by comparing periods of 12 months.

In the data analyses of the impact of shared care the experimental sites are compared with control sites at T1, as well as with all sites at T0, including a difference-in-difference analysis (research questions 4-6). Data analysis on usual health care at T0 will include descriptive analyses and analyses to identify and compare different patient subgroups or patterns of use of health care in this unique combined data set from the several services for a large group of GP patients (research questions 1-2).

SUB-STUDY ON PATIENT-REPORTED HEALTH AND SATISFACTION

Patient-reported mental health, functional impairment due to health problems, overall quality of life and satisfaction with health services are studied for a sub-sample of the register cohort at both T0 and T1. GP patient 16-65 years old are recruited during two weeks at each GP center with some assistance from research staff. Included patients give written consent and complete a brief questionnaire in Norwegian or English. Inclusion criteria and secondary outcome measures in the questionnaire are shown in the tables. The sample is a sub-sample of the register cohorts at T0 and T1. To identify a difference of 6 points on the mental health measure CORE-10 between T0 and T1 with 5% two-tailed significance and 90 % power 70 patients per arm is needed in a cluster randomized trial with ICC=0.03 and 12 GPs in each arm (Eldridge 2012, Schultz 2010, Moher 2010). Aiming to recruit 600-750 patients (20-25 per GP) will secure a more than large enough sub-sample for the main secondary outcome measure (CORE-10). Data analyses of patient-reported information will answer research question 3 and parts of research questions 4 and 5.

QUALITATIVE SUB-STUDY ON EXPERIENCES WITH SHARED CARE

A qualitative sub-study of experiences with collaboration in general, the shared care model, implementation of the model, facilitators and barriers is done at the end of the 18 months period of shared care. Focus groups are conducted with the GPs in each of the GP centers (experimental and control centers), and individual qualitative interviews are done with approximately 15 patients with experience of shared care, nurses and other co-workers at the GP centers, professionals involved with shared care in the primary health and social services, managers at the CMHC and the psychologists and psychiatrist from CMHC working in the shared care. This qualitative study is done in stead of a planned survey with a questionnaire to health personnel, as the number of potential informants would be too small for statistical analyses compared to what was expected when planning the study. Analyses of the qualitative data will answer the research questions 7-9.

ETHICAL APPROVAL

The study protocol was approved by the Regional Committee on Medical and Health Research Ethics Health Region South East 08 May 2014 (reg.no. 2014/435), by the National Committee on Medical and Health Research Ethics in Norway 10 November 2014 (reg.no. 2014/160) and by the Data Protection Officer at Akershus University Hospital (reg.no. 13/138). The National Committee on Medical and Health Research Ethics approved that the study fulfilled the necessary legal criteria to extract structured register data from the services without giving the patients information or asking for written consent. The approved protocol of 2014 is attached to this registration.

PROGRESS AND STATUS OF THE STUDY

Data extraction of the register cohorts was done from the GP electronic patient records in 2015 and 2017, from the mental health services at Akershus University Hospital in 2017-2018 and from the NAV (social/welfare services) in 2017-2018. Data collection from the two clinical cohorts at the GP centers was done in 2015 and 2017. Quality control and organization of data was done 2017-2018. Data analysis starts in September 2018.

ELIGIBILITY:
Inclusion Criteria:

* Seen by a GP during the 12 months for extracted data on all contact

Exclusion Criteria:

* No exclusion criteria

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The total sample of patients seen by any of the GPs at the six participating GP centers during the 12 months of retrospective data extraction from patient registers before randomization of GP centers to shared care, and patients seen by any of the GPs at the six participating GP centers during the 12 months of retrospective data extraction from patient registers during the period where three of the GP centers have shared care. The samples from the two time periods are different, but they may partly overlap as many patients are expected to se GPs during both periods.
Sampling Method: Non-Probability Sample
Enrollment: 19000 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Referrals from GPs to mental health outpatient clinics | 12 months
  Referrals from GPs to mental health outpatient clinics during the period for data extraction

SECONDARY OUTCOMES:
Referrals from GPs to mental health inpatient wards | 12 months
  Referrals from GPs to mental health inpatient wards during the period for data extraction
Waiting time from the referral to the first consultation | 12 months
  Days from the outpatient clinic has received a referral to the first consultation for a referral during the period for data extraction
Number of GP consultations | 12 months
  Number of patient consultations at the GP center during the period for data extraction
Number of outpatient consultations | 12 months
  Number of patient consultations at the outpatient clinic during the period for data extraction
Number of inpatient days | 12 months
  Total number of inpatient days across all inpatient stays during the period for data extraction
Length of an outpatient treatment episode | 12 months
  Days from first consultation to last consultation of a series of outpatient consultations after a referral to the outpatient clinic during the period for data extraction
Length of an inpatient stay | 12 months
  Days from the inpatient admission to discharge after a referral to the inpatient ward during the period for data extraction
Length of sick leave | 12 months
  Days from first to last day of a period of sick leave clinic during the period for data extraction
Type of health problem | 12 months
  ICPC-2 codes in PG practices and/or ICD-10 diagnosis in mental health care during the period for data extraction
The severity of psychiatric symptoms | 12 months
  Global Assessment of Functioning - subscale for symptoms (GAF-S), used in mental health services
The severity of impairment in functioning | 12 months
  Global Assessment of Functioning - subscale for functional impairment (GAF-F), used in mental health services
Self-reported mental health problems | 2 weeks
  In the questionnaire to patients: Clinical Outcome in Routine Evaluation (CORE-10) with 10 items on mental health problems (Barkham 2013). Each item is answered on a 5-point scale of frequency from 0="not at all" to 4="most of the time". The 10 items comprise the following: depression (2 items), anxiety (2 items), functioning (3 items, 1 each for 'general' 'social', and 'close'); trauma (1 item); physical (1 item); and suicidal risk (1 item). Two of the items are positively framed. The ten items are summed (reversing the two positive items) to a total score with a range from 0 to 40, where a higher total sum score means more severe mental health problems.
Self-reported impairment in functioning due to health problems | 2 weeks
  In the questionnaire to patients: Work and Social Adjustment Scale (WSAS) with five items on impairment of functioning in various domains due to health problems (Mundt 2002). Each item is answered on a 5-point scale of degree of impairment from 0="not at all" to 4="very much" (adapted from the original 9-point scale from 0 to 8 to fit with the 5-point scales in the rest of the brief questionnaire). The five items comprise the following: Work/education, housework, social activities, activities alone, contact/relationship with family/others. The five items are summed to a total score with a range from 0 to 20, where a higher total sum score means more severe impairment of functioning due to health problems.
Patient satisfaction with health services | 2 weeks
  In the questionnaire to patients and developed for the study: Three items for a subscale on satisfaction with the GP (for access, met with respect, get help as needed), three items for a subscale on satisfaction with the mental health services (for access, met with respect, get help as needed) if such contact last 12 months, and three items for a subscale on satisfaction with the collaboration between the health services (their collaboration, their understanding of the situation, the usefulness of their total help). Each item is answered on a 5-point scale of degree of impairment from 1="very dissatisfied" to 5="very satisfied". For each subscale the three items are summed to a total score with a range from 3 to 15, where a higher total sum score means a higher degree of satisfaction with the specific services.
Overall quality of life (MANSA) | 2 weeks
  In the questionnaire to patients: A single question on overall quality of life is taken from the Manchester Short Assessment of Quality of Life (MANSA), which is a questionnaire on quality of life used in many recent studies (Priebe 1999). The question is answered on a 5-point scale of degree of satisfaction with overall quality of life from 1="very dissatisfied" to 5="very satisfied" (adapted from the original 7-point scale in MANSA to fit with the 5-point scales in the rest of the brief questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Tormod Fladby, Dr.Med., Study Director — University Hospital, Akershus

REFERENCES:
- [Background] Smith SM, Allwright S, O'Dowd T. Effectiveness of shared care across the interface between primary and specialty care in chronic disease management. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD004910. doi: 10.1002/14651858.CD004910.pub2. PMID 17636778
- [Background] Harkness EF, Bower PJ. On-site mental health workers delivering psychological therapy and psychosocial interventions to patients in primary care: effects on the professional practice of primary care providers. Cochrane Database Syst Rev. 2009 Jan 21;2009(1):CD000532. doi: 10.1002/14651858.CD000532.pub2. PMID 19160181
- [Background] Butler M, Kane RL, McAlpine D, Kathol R, Fu SS, Hagedorn H, Wilt T. Does integrated care improve treatment for depression? A systematic review. J Ambul Care Manage. 2011 Apr-Jun;34(2):113-25. doi: 10.1097/JAC.0b013e31820ef605. PMID 21415610
- [Background] Hviding K, Bugge P, Ekern P, Brelin P, Høifødt TS, Nessa J, Flottorp S (2006). Samhandling om pasienter med alvorlige psykiske problemer i allmennpraksis. [Collaboration regarding patients with severe mental problems in general practice]. Rapport Nr 1-2008. Oslo, Nasjonalt kunnskapssenter for helsetjenesten, 2008.
- [Background] Craven MA, Bland R. Better practices in collaborative mental health care: an analysis of the evidence base. Can J Psychiatry. 2006 May;51(6 Suppl 1):7S-72S. PMID 16786824
- [Background] Kates N, Mazowita G, Lemire F et al (2011a). The Evolution of Collaborative Mental Health Care in Canada; A shared vision for the future. Position paper. The Canadian Journal of Psychiatry 56(5).
- [Background] Kates N, McPherson-Doe C, George L. Integrating mental health services within primary care settings: the Hamilton Family Health Team. J Ambul Care Manage. 2011 Apr-Jun;34(2):174-82. doi: 10.1097/JAC.0b013e31820f6435. PMID 21415615
- [Background] Eldridge S, Kerry S. A practical guide to cluster randomised trials in health services research. John Wiley & Sons, Chichester, UK, 2012
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624
- [Background] Barkham M, Bewick B, Mullin T, Gilbody S, Connell J, Cahill J, Mellor-Clark J, Richards D, Unsworth G, Evans C. The CORE-10: A short measure of psychological distress for routine use in the psychological therapies, Counselling and Psychotherapy Research: Linking research with practice, 2013. 13(1):1-13,
- [Background] Mundt JC, Marks IM, Shear MK, Greist JH. The Work and Social Adjustment Scale: a simple measure of impairment in functioning. Br J Psychiatry. 2002 May;180:461-4. doi: 10.1192/bjp.180.5.461. PMID 11983645
- [Background] Priebe S, Huxley P, Knight S, Evans S. Application and results of the Manchester Short Assessment of Quality of Life (MANSA). Int J Soc Psychiatry. 1999 Spring;45(1):7-12. doi: 10.1177/002076409904500102. PMID 10443245
- [Result] Piiksi Dahli M, Brekke M, Ruud T, Haavet OR. Prevalence and distribution of psychological diagnoses and related frequency of consultations in Norwegian urban general practice. Scand J Prim Health Care. 2020 Jun;38(2):124-131. doi: 10.1080/02813432.2020.1783477. Epub 2020 Jun 27. PMID 32594819
- [Result] Rugkasa J, Tveit OG, Berteig J, Hussain A, Ruud T. Collaborative care for mental health: a qualitative study of the experiences of patients and health professionals. BMC Health Serv Res. 2020 Sep 9;20(1):844. doi: 10.1186/s12913-020-05691-8. PMID 32907559
- [Result] Kann IC, Dahli MP, Ruud T. New collaborative model for patients with mental health problems: Impact on sickness abscence or rehabilitation benefits? [Ny samhandlingsmodell for pasienter med psykiske lidelser: Påvirkes sykefravær eller arbeidsavklaringspenger?] Arbeid og velferd 2019 (2): 27-41
- [Result] Dahli MP, Saltyte-Benth J, Haavet OR, Ruud T, Brekke M. Somatic symptoms and associations with common psychological diagnoses: a retrospective cohort study from Norwegian urban general practice. Fam Pract. 2021 Nov 24;38(6):766-772. doi: 10.1093/fampra/cmab038. PMID 34196347
- [Result] Haavet OR, Saltyte Benth J, Gjelstad S, Hanssen-Bauer K, Dahli MP, Kates N, Ruud T. Detecting young people with mental disorders: a cluster-randomised trial of multidisciplinary health teams at the GP office. BMJ Open. 2021 Dec 24;11(12):e050036. doi: 10.1136/bmjopen-2021-050036. PMID 34952870
- [Result] Tveit OG, Ruud T, Hanssen-Bauer K, Haavet OR, Hussain A. An explorative study of factors associated with treatment in specialized mental health care centers among GP patients in Norway. BMC Health Serv Res. 2021 Sep 13;21(1):960. doi: 10.1186/s12913-021-06982-4. PMID 34517868
- [Result] Dahli MP, Haavet OR, Ruud T, Brekke M. GPs' identification of patients with mental distress: a coupled questionnaire and cohort study from norwegian urban general practice. BMC Prim Care. 2022 Oct 9;23(1):260. doi: 10.1186/s12875-022-01865-x. PMID 36210430

DOCUMENTS (1):
  • Study Protocol (2014-02-12): https://cdn.clinicaltrials.gov/large-docs/29/NCT03624829/Prot_000.pdf